CLINICAL TRIAL: NCT04596579
Title: SARS-CoV-2 Immune Surveillance Among a Population Based Sample of Adults in Florida
Brief Title: SARS-CoV-2 (COVID-19) Immune Surveillance Among a Population Based Sample of Adults in Florida
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-20635
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Coronavirus Infection
Keywords: COVID -19; SARC-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants age 18-34: Up to 300 participants age 18-34 who received an invitation by mail and are free of fever at time of interview.
  Interventions: Diagnostic Test: SARS-CoV-2 Antibody Analysis; Diagnostic Test: Weck-cel Swab Collection; Behavioral: Web Based Questionnaire
- Participants age 35-54: Up to 300 Participants age 35-54 who received an invitation by mail and are free of fever at time of interview.
  Interventions: Diagnostic Test: SARS-CoV-2 Antibody Analysis; Diagnostic Test: Weck-cel Swab Collection; Behavioral: Web Based Questionnaire
- Participants age 55-64: Up to 300 participants age 35-54 who received an invitation by mail and are free of fever at time of interview.
  Interventions: Diagnostic Test: SARS-CoV-2 Antibody Analysis; Diagnostic Test: Weck-cel Swab Collection; Behavioral: Web Based Questionnaire
- Participants 65 and over: Up to 300 participants age 35-54 who received an invitation by mail and are free of fever at time of interview.
  Interventions: Diagnostic Test: SARS-CoV-2 Antibody Analysis; Diagnostic Test: Weck-cel Swab Collection; Behavioral: Web Based Questionnaire

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 Antibody Analysis — 10 ml of blood will be drawn for antibody analysis. Participants who test SARCS-CoV-2 positive will be invited to participate in follow-up antibody testing at 4 weeks and at 3 months.
Diagnostic Test: Weck-cel Swab Collection — A Weck-cel swab will be used to collect secretions from the mucosal epithelium
Behavioral: Web Based Questionnaire — A brief web enabled questionnaire will be administered to collect information related to demographics, SARS-CoV-2 exposure history, past symptoms, comorbidities associates with increased infection and disease risk, as well as immunosuppression status and use to immunosuppressive medications.

SUMMARY:
The overall goal of this study is to understand the immune response (IgG) to SARS-CoV-2 to fill critical knowledge gaps in the natural history of this virus and to inform the development of future infection mitigation efforts. The study team aims to assess the prevalence of circulating IgG antibodies to SARS-CoV-2 and the factors associated with sero-prevalence. These data will be used to estimate the total population that has been exposed to the virus (asymptomatic and symptomatic), the proportion of the population that may be protected by natural immunity, and the proportion that is susceptible. Data obtained from this research will be shared with the Florida Department of Health.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Hillsborough County, Florida
* 18 years of age or older
* Currently not exhibiting symptoms of SARS-CoV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 1135 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who test positive for SARS-CoV-2 antibodies at first visit | At study start
  All participants who respond to study invitation letter will be tested for SARS-CoV-2 antibodies after completing a web-based questionnaire.
Percentage of Participants who test positive for SARS-CoV-2 antibodies at second visit | At 4 weeks
  Participants who tested positive for SARS-CoV-2 antibodies at first study visit will be tested for antibodies to SARS-CoV-2 again at 4 weeks.
Percentage of Participants who test positive for SARS-CoV-2 antibodies at third visit | At 3 months
  Participants who tested positive for SARS-CoV-2 antibodies at second study visit will be tested for antibodies to SARS-CoV-2 again at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anna R Giuliano, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center's Clinical Trials Website — https://moffitt.org/clinical-trials-research/clinical-trials